CLINICAL TRIAL: NCT06624631
Title: Delivery Strategies for Malaria Chemoprevention in the Post-discharge Management of Children Hospitalised With Severe Anaemia or Severe Malaria: Cluster and Individually Randomised Controlled Implementation Trial and Economic Evaluation in Kenya
Brief Title: PDMC Implementation Trial in Kenya
Acronym: PDMC-SL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Institut de Recherche Clinique du Benin (IRCB), Benin (Unknown); Epicentre, Paris, France. (Unknown); Institute of Research for Development, France (Other Government); Training Research Unit of Excellence, Blantyre, Malawi (Unknown); Makerere University (Other); Centres for Disease Control and Prevention, Kenya. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-023
Record Dates: First submitted 2024-08-01; First posted 2024-10-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Severe Malaria; Severe Anemia
Keywords: Children; Antimalarial; Prevention; Chemoprevention; Caregivers; Patient discharge; Healthcare providers; Health economics; Qualitative research; Feasibility; Cost effectiveness; Kenya; Artemisinins; School age; Pre-school
MeSH Terms: conditions — Malaria; Anemia | interventions — somatostatin, cyclic hexapeptide(Phe-Phe-Trp-Lys-Thr-Phe)-; House Calls

STUDY DESIGN:
Intervention Model Description: A multi-centre, 2-arm, cluster-randomised trial evaluating two health system delivery strategies and a 3-arm nested individually randomised trial evaluating two new intervention strategies to enhance end-user adherence to post-discharge malaria chemoprevention (PDMC) with dihydroartemisinin-piperaquine compared to the standard of care without adherence strategies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decentralized, monthly delivery of Post Discharge Malaria Chemoprevention (PDMC) drugs (Arm A) (Experimental): Delivery of initial course of PDMC at discharge from the admitting facility. Referral to caregiver's peripheral facility of choice for delivery of subsequent monthly courses
  Interventions: Other: SMS reminders; adherence support strategy a; Other: Community Health Promoters (CHP) home visits; adherence support strategy b; Other: No reminders; adherence support strategy c
- Centralised delivery of Post Discharge Malaria Chemoprevention (PDMC) drugs at discharge (Arm B) (Active Comparator): Delivery of all three courses of Post Discharge Malaria Chemoprevention (PDMC) drugs at discharge from the admitting facility.
  Interventions: Other: SMS reminders; adherence support strategy a; Other: Community Health Promoters (CHP) home visits; adherence support strategy b; Other: No reminders; adherence support strategy c

INTERVENTIONS:
Other: SMS reminders; adherence support strategy a — Monthly SMS reminders sent to participants allocated to this adherence support intervention in both drug delivery arms (Centralized and decentralized arms)
Other: Community Health Promoters (CHP) home visits; adherence support strategy b — Community Health Promoters' (CHPs) monthly reminder home visits conducted for participants allocated to this adherence support intervention in both drug delivery arms (Centralized and Decentralized arms)
Other: No reminders; adherence support strategy c — No monthly reminders sent for participants allocated to this control adherence support intervention group in both drug delivery arms (Centralized and Decentralized arms)

SUMMARY:
The goal of this implementation trial is to evaluate at least two alternative delivery strategies and adherence support for malaria chemoprevention with dihydroartemisinin-piperaquine in the post-discharge management of children hospitalised with severe anaemia or severe malaria to optimise adherence in Kenya.

The actual interventions to be evaluated have been co-designed with national stakeholders during an initial formative research stage.

DETAILED DESCRIPTION:
Study design:

A multi-centre, 2-arm, cluster-randomised trial evaluating two health system delivery strategies and a 3-arm nested individually randomised trial evaluating two new intervention strategies to enhance end-user adherence to post discharge malaria chemoprevention (PDMC) with dihydroartemisinin-piperaquine compared to the standard of care without adherence strategies.

Study sites: Health facilities with blood transfusion services in malaria-endemic areas in western Kenya.

Study Population:

Cluster inclusion criteria: health facilities with blood transfusion services offering in-patient care for children with severe anaemia and severe malaria. Exclusion criteria: primary health facilities without subservient lower-level health facilities.

Individual inclusion criteria: convalescent children aged <10 years, weighing ≥5 kg admitted with severe anaemia (haemoglobin<5g/dL) or severe malaria; clinically stable, able to take or switch to oral medication; post-transfusion Hb >5g/dL. Exclusion criteria: blood loss due to trauma, malignancy, known bleeding disorders or sickle cell disease, known hypersensitivity to study drug, known heart conditions, non-resident in the study area, previous participation in the study, known need at enrolment for prohibited medication and scheduled surgery during the 4-month course of the study. HIV infection and cotrimoxazole prophylaxis are not exclusion criteria.

Study Interventions:

Cluster randomised trial: Hospitals will be randomised to one of two delivery platforms for PDMC (A or B). In delivery platform A, the initial course of PDMC will be delivered at discharge at the admitting facility. Subsequent courses will be dispensed during monthly visits to the health facility of their choice.In strategy B, all 3 courses will be dispensed at discharge.

Individually randomised trial: Three different adherence support strategies, including: SMS reminders to caregivers (arm a), Community Health Promoter (CHP) support through home visits (arm b), and a control arm comprising of no additional adherence support (arm c).

All participating children will receive standard in-hospital care for severe anaemia or severe malaria (blood transfusion, often combined parenteral artesunate, followed by a 3-day course of AL (whether they initially had malaria or not), which will be started in-hospital as soon as they are able to take oral medication. Many children are likely to receive parenteral antibiotics as well as part of the standard of care.

Primary endpoints:

Cluster randomised trial: The proportion of eligible participants who were not prescribed the full 3 courses of PDMC.

Individually randomised trial: The proportion of children with incomplete adherence to the 9 doses of PDMC (three courses of 3-day treatments 3x3=9).

Secondary endpoints:

1. Clinical effectiveness (all-cause and malaria-specific sick-child clinic visits, all-cause and cause-specific readmissions and all-cause mortality by the end of week 14 after discharge.
2. Safety (incidence of serious adverse events).
3. Cost-effectiveness.
4. Acceptability and feasibility.

Follow-up procedures:

Children will be followed for 14 weeks (i.e., four weeks after the last PDMC course) through passive surveillance of clinic visits and hospitalisations. Each child will then be seen for an end-of-study visit towards the end of week 14. Children will also be visited at home for unannounced home visits one to three days from the last day of the last dose of each 3-day course of PDMC medication to assess adherence.

Sample size:

Cluster randomised trial: A sample size of 51 participants with complete follow-up recruited in 5 control and 5 intervention clusters (300 per arm) provides over 80% power to detect a risk difference of 20% from 35% in the control arm to 15% in the intervention clusters (RR=0.43), using a two-sided alpha of 0.05, and assuming an intra-cluster correlation coefficient (ICC) of 0.03,a coefficient of variation of 0.39 and a small-sample correction at the analysis stage, thus the t-distribution is assumed implying an adjustment in the degrees of freedom. Similarly, the same size would provide over 90% power to detect a risk difference of 23% from 35.0% to 12% (alpha = 0.05) (RR=0.34). To allow for a 15% loss to follow-up and enough power at the individual-level, we aim to recruit approximately 60 participants per cluster, or approximately 600 participants (300 per arm).

Individually randomised trial: A sample size of 147 participants in the control arm (c) and 147 in each of the two intervention arms (a and b), totalling 441 participants, would provide 90% power to detect a 50% reduction in the primary endpoint (proportion of children with incomplete adherence to the 9 doses of PDMC) from 36.8% in the control arm to 18.4% (RR=0.50) in any of the two intervention arms using a 1:1:1 allocation after accounting for the multiple comparisons (α = 0.025). A total of 519 participants (173 per arm) will be recruited to allow for a 15% loss to follow-up.

Data Analysis:

Risk ratios and corresponding 95% confidence intervals will be computed to compare treatment effects using multi-level mixed models accounting for clustering effects.

ELIGIBILITY:
Inclusion Criteria:

CLUSTERS

* Health facilities with blood transfusion services offering in-patient care for children with severe anaemia and severe malaria.
* >=40 children per year admitted with severe anaemia or severe malaria
* Agreement to participate by facility management
* Located in areas with moderate to high malaria transmission

INDIVIDUAL PARTICIPANTS

* Aged <10 years of both sexes
* Hospitalised with severe anaemia or severe malaria: Initially hospitalised with haemoglobin <5.0 g/dl or PCV <15%, or requirement for blood transfusion for other clinical reasons on or during admission to the hospital, or severe malaria, defined as a requirement for parenteral artesunate in the opinion of the treating clinician and/or the presence of microscopy or RDT confirmed Plasmodium infection

Exclusion Criteria:

CLUSTERS

- Health facilities without subservient lower-level health facilities

INDIVIDUAL PARTICIPANTS

* Recognised specific other causes of severe anaemia (i.e., trauma, haematological malignancy, known bleeding disorders, such as haemophilia)
* Sickle cell anaemia/sickle cell disease
* Body weight <5 kg
* HIV infection and cotrimoxazole prophylaxis are not exclusion criteria.

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible children who received 3 courses of PDMC | 2, 6 and 10 weeks post discharge
  Proportion of eligible participants who received all 3 indicated PDMC courses from Ministry of Health staff
Proportion of study children who adhered to 3 PDMC courses (9 doses) | 2, 6 and 10 weeks (days 1-3) post discharge
  Proportion of children with complete adherence to the full PDMC regimen (3 courses × 3 doses = 9 total doses)

SECONDARY OUTCOMES:
Proportion of children who are readmitted with malaria | 0-14 weeks post discharge
  All-cause and malaria-specific sick-child clinic visits by the end of week 14 after discharge
Proportion of children who are readmitted with any cause | 0-14 weeks post discharge
  All-cause and cause-specific readmissions by the end of week 14 after discharge
Proportion of children who die within 14 weeks of discharge | 0-14 weeks post discharge
  All-cause mortality by the end of week 14 after discharge
Incidence of serious adverse events | 0-14 weeks post discharge
  Incidence of serious adverse events
Cost-effectiveness | 0-14 weeks post discharge
  Incremental cost per DALY averted of alternative PDMC adherence support strategies (adherence support option A [Aa], adherence support option B [Ab]) with no adherence support (Ac), and with each other
User and provider perceptions of acceptability and feasibility | Trial month 6+
  Acceptability and feasibility of PDMC delivery strategies

CONTACTS AND LOCATIONS:
Overall Officials: Feiko ter Kuile, MD, PhD, Principal Investigator — LSTM
Locations (1):
- Kemri, Cghr, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared once the publication is accepted by a journal.
Access Criteria: Applications to access data are assessed as per the choice of the data contributor, either by:
  1. An independent IDDO Data Access Committee (DAC)
  2. A contributor-controlled process - where the data contributor assesses each data access application that requests the re-use of their data
URL: http://www.iddo.org/data-sharing/contributing-data